CLINICAL TRIAL: NCT01255722
Title: Xenetix® 350: Comparative Assessment of Image Quality for Coronary CT Angiography (X-ACT Study)
Brief Title: Xenetix® 350: Comparative Assessment of Image Quality for Coronary CT Angiography
Acronym: X-ACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: ISO-44-012
Record Dates: First submitted 2010-12-03; First posted 2010-12-07 (Estimated); Results first posted 2015-12-16 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-11

CONDITIONS: Coronary Artery Disease
Keywords: iodinated contrast media, coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — iobitridol; iopromide; iomeprol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Iobitridol (Experimental): Patients were IV injected with a single dose of iobitridol before a coronary CT angiography
  Interventions: Drug: iobitridol
- Iopromide (Active Comparator): Patients were IV injected with a single dose of iopromide before a coronary CT angiography
  Interventions: Drug: iopromide
- Iomeprol (Active Comparator): Patients were IV injected with a single dose of iomeprol before a coronary CT angiography
  Interventions: Drug: iomeprol

INTERVENTIONS:
Drug: iobitridol — single IV injection
  Other Names: Xenetix®
  Arms: Iobitridol
Drug: iopromide — Single IV injection
  Other Names: Ultravist®
  Arms: Iopromide
Drug: iomeprol — Single IV injection
  Other Names: Iomeron®
  Arms: Iomeprol

SUMMARY:
The purpose of this study is to demonstrate the (statistical) non-inferiority of iobitridol (Xenetix® 350) when compared to contrast agents with higher iodine concentrations, iopromide (Ultravist® 370) and iomeprol (Iomeron® 400) in terms of coronary CT scan evaluability (quality and interpretability of images).

DETAILED DESCRIPTION:
Patients suspected of coronary artery disease were submitted to coronary CT angiography using either iobitridol or contrast agents with higher iodine concentrations (iopromide or iomeprol). Independent off-site readers evaluated image quality regarding the ability to identify coronary artery stenosis (score 0- non evaluable to 4- excellent quality). The study was aimed at showing the non-inferiority of iobitridol in its ability to provide evaluable CT scans for the identification of coronary stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult patient (having reached legal majority age)
* Symptomatic patient suspected for coronary artery disease scheduled for a coronary CT angiography

Exclusion Criteria:

* Patient with a heart rate > 65 beats per minute (bpm) and contraindication or intolerance to b-blocker administration
* Patient with arrhythmia or non-sinus rhythm
* Patient with decompensated heart failure
* Patient with evidence of ongoing or active clinical instability (suspected or known acute myocardial infarction, cardiac shock, acute pulmonary oedema)
* Patient who has previously undergone coronary artery bypass graft
* Patient who has previously undergone percutaneous transluminal coronary stent placement
* Patient with artificial heart valve
* Patient with known moderate to severe aortic stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2010-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin HOFFMANN, MD, Principal Investigator — Kantonsspital Lucerne- Switzerland
Locations (23):
- France (9):
  - CHU Angers, Angers
  - CHU de la Cavale Blanche, Brest
  - Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson
  - La Timone Adultes, Marseille
  - Hopital Cochin, Paris
  - Haut-Lévêque / Radiologie, Pessac
  - CHU Pontchaillou, Rennes
  - CHU Rouen - Hopital Charles Nicolle, Rouen
  - Centre Cardiologique du Nord, Saint-Denis
- Germany (6):
  - Institut für Radiologie Universitätsklinikum Charité, Berlin
  - University Hospital Erlangen, Erlangen
  - Elisabeth-Krankenhaus Hospital, Essen
  - University Hospital Mannheim, Mannheim
  - University Hospital LMU, Munich
  - Universitätsklinik Ulm, Ulm
- Italy (4):
  - Ospedale A.Perrino U.O. di radiodiagnostica, Brindisi
  - Ospedale del Delta, Ferrara
  - Sapienza-universita di Roma, Rome
  - Ospedale civile Maggiore du Verona Borgo, Verona
- Spain (3):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Complejo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela
- Institut für Radiologie, Sankt Gallen, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 468 patients from 5 European countries were enrolled and evaluated between 3 November 2010 and 17 September 2012.
Period: Overall Study
Arm/Group | Iobitridol | Iopromide | Iomeprol
Started | 155 | 160 | 153
Completed | 152 | 159 | 152
Not Completed | 3 | 1 | 1
Not completed — Adverse Event | 0 | 1 | 1
Not completed — asymptomatic patient | 1 | 0 | 0
Not completed — beta-blocker contraindicated | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All included patients set: all included patients, even those who have withdrew prior to contrast injection.
Groups:
- Total: Total of all reporting groups
Arm/Group | Iobitridol | Iopromide | Iomeprol | Total
Number analyzed (Participants) | 155 | 160 | 153 | 468
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 104 | 101 | 108 | 313
  >=65 years | 51 | 59 | 45 | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (12.2) | 58.7 (11.6) | 56.9 (13.4) | 57.8 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 68 | 65 | 198
  Male | 90 | 92 | 88 | 270
Region of Enrollment [Number; unit: participants]
  France | 59 | 61 | 59 | 179
  Spain | 21 | 21 | 20 | 62
  Germany | 41 | 45 | 41 | 127
  Switzerland | 9 | 9 | 10 | 28
  Italy | 25 | 24 | 23 | 72

OUTCOME MEASURES:

1. Primary Outcome: Rate of Patients With Evaluable CT Scans i.e. Allowing Identification of Coronary Artery Stenosis According to Off-site Reading Assessment
Description: Evaluability was based upon the off-site assessment of 18-coronary segments graded for image quality with a 5-point scale.4= Excellent quality, fully confidence without any doubts concerning the presence/absence of luminal stenosis; 3= Good quality, confidence concerning the presence/absence of luminal stenosis; 2= Moderate quality, relative confidence, with minor doubts concerning the presence/absence of luminal stenosis; 1= Poor quality, some doubts concerning the presence/absence of stenosis; 0= Non diagnostic.
  A patient's CT scan was considered as evaluable for identification of coronary artery stenosis if none of the 18 coronary segments had a score of 0.
Time Frame: < 24h
Population: Full Analysis Set: all patients who underwent the coronary CT scan examination and had available assessments of the primary endpoint.
Measure: Geometric Mean (Standard Error); unit: Percentage of patients
Arm/Group | Iobitridol | Iopromide | Iomeprol
Number analyzed (Participants) | 151 | 152 | 149
Percentage of patients | 92.1 (2.2) | 95.4 (1.7) | 94.6 (1.8)
Statistical Analysis 1: Comparison: Iobitridol vs Iopromide vs Iomeprol; Iobitridol was compared to the best of the two comparators. The two-sided 95% confidence interval (CI) of the difference between both proportions (Iobitridol - Comparator) was computed and the lower limit of the CI compared to the clinical non-inferiority limit in the study. The non-inferiority of iobitridol over the best comparator was established if the lower limit of the two-sided 95% CI was equal to or higher than the clinical non-inferiority limit; Test type: Non-Inferiority or Equivalence — The clinical non-inferiority margin was set to -10% maximum difference with the best comparator (i.e. iopromide); p = 0.05, Chi-squared; Mean Difference (Final Values) = -0.033, 95% CI 2-sided [-0.088 to 0.021]

2. Secondary Outcome: Average Image Quality According to Off-site Reading
Description: For each patient, all 18 coronary segments were graded for image quality using a 5-point evaluation scale (from 0=non-diagnostic to 4=excellent). The average image quality was evaluated using the off-site readings, by averaging the scores obtained for the 18 segments used to determine the CT evaluability (primary criteria).
Time Frame: <24h
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Image quality Score on a scale
Groups:
- Iopromide: Patients were IV injected with a single dose of iopromide before coronary CT angiography
Arm/Group | Iobitridol | Iopromide | Iomeprol
Number analyzed (Participants) | 151 | 152 | 149
Image quality Score on a scale | 3.5 (0.9) | 3.5 (0.8) | 3.4 (0.9)
Statistical Analysis 1: Comparison: Iobitridol vs Iopromide vs Iomeprol; Test type: Superiority or Other; p = 0.750, Fisher Exact

3. Secondary Outcome: Coronary Track Rate
Description: A post processing software automatically tracked the number of distal segments of the left anterior descending coronary artery, the left circumflex coronary artery and the right coronary artery . The number of segments tracked per patient were assessed by an independent off-site radiologist.
Time Frame: <24h
Population: Full Analysis Set population: all patients who underwent the coronary CT scan examination and had available assessments of the primary endpoint.
Measure: Mean (Standard Deviation); unit: Number of tracked segments per patient
Arm/Group | Iobitridol | Iopromide | Iomeprol
Number analyzed (Participants) | 151 | 152 | 149
Number of tracked segments per patient | 10.9 (2.2) | 10.8 (2.4) | 11.1 (2.3)

4. Secondary Outcome: Average Signal Attenuation After IV Injection of Contrast
Description: Attenuation of signal was measured off-site on post-injection images of four coronary segments, in the ascending aorta and in the left ventricle, then it was averaged at the patient level.
Time Frame: <1h
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: Hounsfield Units
Arm/Group | Iobitridol | Iopromide | Iomeprol
Number analyzed (Participants) | 151 | 152 | 149
Hounsfield Units | 426.3 (92.9) | 449.8 (88.1) | 466.4 (104.6)
Statistical Analysis 1: Comparison: Iobitridol vs Iopromide vs Iomeprol; Test type: Superiority or Other; p = 0.001, Fisher Exact

5. Secondary Outcome: Average Signal-to-Noise Ratio (Average SNR)
Description: Signal attenuation was measured by off-site radiologists in the lumen of 4 coronary segments, in the ascending aorta and in the left ventricle and was expressed in Hounsfield Unit (HU). Measurements were set in post-injection images for the 6 territories.
  A measure of noise in CT scans was collected at least in the aorta and if possible in the muscle and/or air.
  Signal-to-Noise Ratios (SNR) of post-injection images were derived in all territories from attenuation measurements according to the following formula:
  SNR Territory = Post Attenuation / Image Noise
Time Frame: <1h
Population: Full Analysis Set: included all patients who underwent the examination and had available assessments of the primary endpoint.
Measure: Mean (Standard Deviation); unit: Hounsfield Units:Hounsfield Units
Arm/Group | Iobitridol | Iopromide | Iomeprol
Number analyzed (Participants) | 151 | 152 | 149
Hounsfield Units:Hounsfield Units | 16.2 (5.6) | 17.1 (5.0) | 17.6 (6.6)
Statistical Analysis 1: Comparison: Iobitridol vs Iopromide vs Iomeprol; Test type: Superiority or Other; p = 0.109, Fisher Exact

6. Secondary Outcome: Average Contrast-to-noise Ratio (Average CNR)
Description: Signal attenuation was measured by off-site radiologists in the lumen of 4 coronary segments in the ascending aorta and the in left ventricle and expressed in Hounsfield Unit (HU).
  A measure of noise in CT scans was collected at least in the aorta and if possible in the muscle and/or air.
  In territories where pre and post signal attenuation measures were both available, the contrast-to-noise ratio was computed according to the following formula: CNR = (Post Att - Baseline Att) / Image Noise
Time Frame: <1h
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Hounsfield Units:Hounsfield Units
Arm/Group | Iobitridol | Iopromide | Iomeprol
Number analyzed (Participants) | 151 | 152 | 149
Hounsfield Units:Hounsfield Units | 14.4 (5.4) | 15.3 (4.8) | 15.8 (6.5)
Statistical Analysis 1: Comparison: Iobitridol vs Iopromide vs Iomeprol; Test type: Superiority or Other; p = 0.09, Fisher Exact

ADVERSE EVENTS:
Time Frame: Post-injection adverse events (i.e. treatment-emergent adverse events) were reported from the time of injection of the contrast media up to 30 minutes after the end of the CT scan exam.
Description: The Official French Method of Causality Assessment was used (Begaud B et al. 'Imputation of the unexpected or toxic effects of drugs. Actualization of the method used in France'. Therapy. 1985;40:111-8).
Arm/Group | Iobitridol | Iopromide | Iomeprol
Serious Adverse Events (participants affected / at risk) | 0/152 | 0/159 | 1/152
Other Adverse Events (participants affected / at risk) | 23/152 | 31/159 | 23/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iobitridol (N=152) | Iopromide (N=159) | Iomeprol (N=152)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iobitridol (N=152) | Iopromide (N=159) | Iomeprol (N=152)
Bradycardia (Cardiac disorders) | 11 (12) | 16 (17) | 12 (13)
Extrasystoles (Cardiac disorders) | 11 (11) | 7 (8) | 7 (7)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3)
Injection Site Pain (General disorders) | 0 (0) | 3 (3) | 2 (2)
Pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Arrythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The main limitation of the study is the absence of gold standard such as conventional angiography to confirm the readers' assessments. Diagnostic accuracy could therefore not be compared.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished data given to the investigator may be transmitted to a third party without prior approval of the sponsor in writing. The data are the exclusive property of Guerbet.

The investigator undertakes to submit to Guerbet any draft articles or papers related to this study within 30 days of their submission to the scientific review or the congress scientific committee.

All written or oral papers and publications must have the joint agreement of the investigator and the sponsor.